CLINICAL TRIAL: NCT05725889
Title: Detection of Visual-Auditory Reaction Rates in Individuals With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, melisa bilaloğlu, RESEARCH ASSISTANT, Baskent University
Other Study IDs: 193.140.162.4
Record Dates: First submitted 2022-11-29; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Dysfunction; Nerve Damage
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DIABETES: Visual, finger tapping and auditory tests were performed regularly. The subjects' fasting plasma glucose and HbA1c levels, and the duration of their diabetes were recorded.
  Interventions: Device: recation time test
- CONTROL: Visual, finger tapping and auditory tests were performed regularly. The subjects' fasting plasma glucose and HbA1c levels were recorded.
  Interventions: Device: recation time test

INTERVENTIONS:
Device: recation time test — visual-finger tapping and auditory reaction time tests

SUMMARY:
Background: The primary purpose of our study was to understand the damage in the peripheral nerves of patients with diabetes and to determine the change in patients' reaction rates and perceptions by the age groups, duration of diabetes, fasting plasma glucose and HbA1c values, and compare these with those of the healthy individuals.

Methods: This study was carried out at the Baskent University Hospital Endocrinology and Metabolic Diseases Outpatient Clinic. A total of 64 patients diagnosed with type 2 diabetes and 64 healthy controls were included in the study. Finger tapping, visual, and auditory reaction time tests were performed on the subjects, respectively. The subjects' fasting plasma glucose and HbA1c levels, and the duration of their diabetes were recorded. Analyses were performed using the SPSS version 25. Differences were considered statistically significant when the p-value is <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed individuals
* Must be between 18-65 ages
* Must be Type 2 diabetics at least 6 months (for patient group)

Exclusion Criteria:

* use of alcohol-drug or similar substances,
* the use of any medication that may affect neurological functions,
* having color blindness,
* retinopathy,
* neurological disease,
* cancer,
* depression,
* a recent history of surgery,
* rheumatoid arthritis,
* osteoarthritis,
* and advanced osteoarthritis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consisted of healthy individuals aged between 18-64 years, diagnosed with type 2 diabetes, and resided in Ankara. The sample comprised 128 volunteers, 64 of whom were patients and 64 were controls.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Finger tap, visual and auditory reaction test data within 10 seconds | April-September 2021
  Reaction times

CONTACTS AND LOCATIONS:
Overall Officials: melisa bilaloğlu, res asst, Study Chair — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided